CLINICAL TRIAL: NCT02364583
Title: Safety, Tolerability and Pilot Efficacy of Short Course, High Dose Primaquine Treatment for Liver Stages of Plasmodium Vivax Infection
Brief Title: Investigation of Short Course, High Dose Primaquine Treatment for Liver Stages of Plasmodium Vivax Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); The University of Western Australia (Other); University of Oxford (Other); Curtin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRAC10.14
Record Dates: First submitted 2014-11-13; First posted 2015-02-18 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Plasmodium Vivax
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 14 day dose regimen (Active Comparator): 0.5 mg/kg oral Primaquine administered daily for 14 days
  Interventions: Drug: Primaquine
- 7 day dose regimen (Active Comparator): 1.0 mg/kg oral Primaquine administered daily for 7 days
  Interventions: Drug: Primaquine
- 3.5 day dose regimen (Active Comparator): 1.0 mg/kg oral Primaquine administered twice daily (bd) for 3.5 days
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Primaquine treatment given in a step-wise manner; (a) 0.5 mg/kg total dose daily for 14 days (n=40), (b) 1.0 mg/kg total dose daily for 7 days (n=40), (c) 1.0 mg/kg twice daily for 3.5 days (n=40)
  Other Names: Primaquine phosphate

SUMMARY:
This study specifically seeks to provide data on the safety, tolerability and pilot efficacy of short course, high dose primaquine treatment in Papua New Guinean children aged 5-10 years, in a cross-sectional study design. Community screened asymptomatic cases and/or cases of clinically diagnosed malaria admitted to the out-patient units of the health center, will be screened for Glucose-6-phosphate dehydrogenase deficiency (G6PD) and malaria illness by rapid diagnostic test and P. vivax infection confirmed by light microscopy. Following treatment with artemether-lumefantrine (Coartem), G6PD normal children will be enrolled into the study and followed for 2 months. Primaquine treatment will be allocated to study participants in a step-wise design; firstly receiving the current 14 day treatment regimen of 0.5 mg/kg total dose (n=40); secondly, a 7 day treatment regimen receiving a total dose of 1.0 mg/kg/day; then thirdly, receive 1.0 mg/kg twice daily dose (bd) for a total of 3.5 days, should the 7 day treatment prove to be safe and well tolerated. In addition to this dose-escalation study, the pharmacokinetic profiles of single doses of 0.5 mg/kg and 1.0 mg/kg will be determined using an intensive sampling protocol, in children aged 5-10 years. The pharmacokinetic profiles obtained by this sub-study will be essential for modeling the population pharmacokinetic data obtained from the dose-escalation study. As there is currently no data on the safety, tolerability and efficacy of primaquine in children, the present study will validate previous observation and contribute to the knowledge of primaquine as a treatment for liver stages of Plasmodium vivax infection.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident in study area
* Absence of history of hypersensitivity reactions to pre-treatment drugs
* Positive for P. vivax infections on blood smear or PCR
* Normal G6PD enzyme activity

Exclusion Criteria:

* Features of severe malaria
* Clinical evidence of nonmalarial illness
* Severe malnutrition (weight for age nutritional Z score <60th percentile)
* Moderate to severe anemia (Hb <8g/dL)
* Permanent disability which prevents or impedes study participation

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by hemoglobin | 2 months post baseline
Safety and tolerability as measured by methemoglobin | 2 months post baseline
Safety and tolerability as measured by liver biochemistry | 2 months post baseline
Safety and tolerability as measured by symptom questionnaire | 2 months post baseline

SECONDARY OUTCOMES:
Time to first or only Plasmodium vivax infection by light microscopy and polymerase chain reaction (PCR) | 2 months from baseline
  Thick and thin blood films, along with PCR samples, will be collected at time of recruitment and then at any time the participant develops fever within the study period.
Time to first or only clinical Plasmodium vivax episode | 2 months from baseline
Comparison of the rate of incidence of P. vivax relapses in 3.5 or 7 day treatment arm compared to standard 14 day regimen | 2 months from baseline
Pharmacokinetics - elimination half-life (t1/2) | 42 days
Pharmacokinetics - clearance (CL) | 42 days
Pharmacokinetics - volume of distribution (Vd) | 42 days
Pharmacokinetics - maximal concentration (Cmax) | 42 days
Pharmacokinetics - area under the curve (AUC) | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Inoni Betuela, MD, PhD, Principal Investigator — PNG Institute of Medical Research; Ivo Mueller, PhD, Principal Investigator — Walter and Eliza Hall Institute of Medical Research; Centre de Recerca en Salut Internacional de Barcelona (CRESIB); J Kevin Baird, PhD, Principal Investigator — Eijkman-Oxford Clinical Research Unit, Oxford University; Timothy ME Davis, FRAC, PhD, Principal Investigator — The University of Western Australia
Locations (1):
- PNG Institute of Medical Research, Madang, Madang Province, Papua New Guinea

REFERENCES:
- [Derived] Moore BR, Salman S, Tobe R, Benjamin J, Yadi G, Kasian B, Laman M, Robinson LJ, Page-Sharp M, Betuela I, Batty KT, Manning L, Mueller I, Davis TME. Short-course, high-dose primaquine regimens for the treatment of liver-stage vivax malaria in children. Int J Infect Dis. 2023 Sep;134:114-122. doi: 10.1016/j.ijid.2023.05.063. Epub 2023 Jun 1. PMID 37269941